CLINICAL TRIAL: NCT01263743
Title: Relaxation Response Training to Treat Hypertension: Effects on Blood Pressure, Biomarkers, and Endothelial Function
Brief Title: Relaxation Response Training to Treat Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jeff C. Huffman, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2008P002244
Record Dates: First submitted 2010-12-14; First posted 2010-12-21 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Hypertension
Keywords: Stage 1 hypertension
MeSH Terms: conditions — Hypertension | interventions — Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- This is a single arm study (Experimental): Relaxation Response training will be given to all participants
  Interventions: Behavioral: Relaxation Response

INTERVENTIONS:
Behavioral: Relaxation Response — The Relaxation Response is a type of relaxation. The goal of the Relaxation Response is to consciously elicit a reaction opposite in direction to the stress response.
  Other Names: Meditation
Behavioral: Relaxation Response — Relaxation Response is a type of relaxation. This is a technique that elicits a state that is opposite to the stress response.
  Other Names: Meditation

SUMMARY:
Interventions such as Relaxation Response appear to have widespread effects on physiology. Endothelial function, changes in genomic expression, several biomarkers have been associated with chronic stress and cardiovascular dysfunction, and there is some suggestion that elicitation of the Relaxation Response may lead to improvement in-or normalization of-these factors. By studying the impact of the Relaxation Response on endothelial function, genomic expression and biomarkers among subjects with hypertension, it may be possible to better understand the biologic underpinnings of Relaxation Response-type interventions. Furthermore, with a greater understanding of the physiologic mechanisms by which the Relaxation Response works, it may be possible to better target other symptoms and conditions that can be effectively treated by such an intervention.

ELIGIBILITY:
General Inclusion Criteria:

* Healthy men and women
* Hypertension (stage 1)
* 18-70 years old

General Exclusion Criteria

* No asthma or nasal allergies
* Non-smokers
* If on anti-hypertensive medication willing to discontinue
* Cannot currently practice Tai Chi, meditation, or yoga regularly
* Current use of the following medications: phosphodiesterase type 5 inhibitors, long-acting nitrates, systemic corticosteroids, anti-inflammatories, immunosuppressive or cytotoxic therapies (currently or within the last 12 months), anabolic steroids, and antidepressants.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Endothelial Function | Eight weeks of Relaxation Response Training

SECONDARY OUTCOMES:
Blood Pressure | Eight Weeks of Relaxation Response Training
Genomic Expression | Eight Weeks of Relaxation Response Training

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Huffman, MD, Principal Investigator — Massachusetts General Hospital; Randall Zusman, MD, Study Director — Massachusetts General Hospital; Mark A Creager, MD, Study Director — Brigham and Women's Hospital; John W Denninger, MD, Study Director — Massachusetts General Hospital; Herbert Benson, MD, Study Director — Massachusetts General Hospital; Gregory Fricchione, MD, Study Director — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States